## **SUMMARY OF CHANGES – Consent**

NCI Protocol #: 10250

**Local Protocol #:** 201910106

**Protocol Version Date:** July 12, 2023

Protocol Title: A Phase II Study of the PARP Inhibitor Olaparib in Combination with the DNA

Damaging Agent Temozolomide for the Treatment of Advanced Uterine Leiomyosarcoma

**Informed Consent Version Date:** July 12, 2023

## I. Changes:

| # | Section | Comments |
|---|---|---|
| 1. | Footers | The protocol and informed consent version date was updated to be |
| | | July 12, 2023. |
| 2. | Possible Side | Added New Risk: |
| | Effects of Olaparib | Rare: Blood clot |

Protocol Version Date: July 12, 2023 Page i of i

## **Research Study Informed Consent Document**

Study Title for Participants: A phase II clinical trial evaluating the combination of olaparib and temozolomide for the treatment of advanced uterine leiomyosarcoma

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: Protocol P10250, A Phase II Study of the PARP Inhibitor Olaparib in Combination with the DNA Damaging Agent Temozolomide for the Treatment of Advanced Uterine Leiomyosarcoma (NCT#: 03880019)

## **Overview and Key Information**

## What am I being asked to do?

We are asking you to take part in a research study. This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

We are asking you to take part in this research study because you have been diagnosed with advanced uterine leiomyosarcoma (LMS).

## Taking part in this study is your choice.

You can choose to take part or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document has important information to help you make your choice. Take time to read it. Talk to your doctor, family, or friends about the risks and benefits of taking part in the study. It's important that you have as much information as you need and that all your questions are answered. See the "Where can I get more information?" section for resources for more clinical trials and general cancer information.

# Why is this study being done?

This study is being done to answer the following question:

Will the combination of olaparib and temozolomide be a safe and effective treatment for patients with advanced uterine leiomyosarcoma after at least one prior treatment for the cancer has stopped working?

We are doing this study because we want to find out if this approach is better or worse than the usual approach for uterine leiomyosarcoma after at least one prior treatment has stopped


working. The usual approach is defined as care most people get for uterine leiomyosarcoma in this situation.

## What is the usual approach to my uterine leiomyosarcoma?

The usual approach for patients with advanced uterine leiomyosarcoma who are not in a study will include treatment with a drug that is approved by the Food and Drug Administration (FDA) for the treatment of this disease. These drugs include systemic chemotherapy, such as: doxorubicin (alone or in combination with ifosfamide), gemcitabine and docetaxel, trabectedin, or dacarbazine. Patients might also receive pazopanib, an oral targeted drug, which is usually used after chemotherapy stops working or causes too many side effects. The decision about which of these drugs is best would be made by your oncologist after consulting with you.

## What are my choices if I decide not to take part in this study?

- You may choose to have the usual approach described above.
- You may choose to take part in a different research study, if one is available.
- You may choose not to be treated for cancer.
- You may choose to only receive comfort care to help relieve your symptoms and not be treated for your cancer.

## What will happen if I decide to take part in this study?

If you decide to take part in this study, you will receive olaparib and temozolomide for as long as this treatment is helping you and not causing side effects that are too severe.

After you finish the olaparib and temozolomide treatment, your doctor will continue to follow your condition and watch you for side effects. Your doctor may follow-up with you by phone call every 3 months for a period of up to 2 years after the study ends. The study team may continue to contact you every 6 months after this period to ask about specific side effects from the treatment.

# What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision.

#### **Risks**

We want to make sure you know about a few key risks right now. We give you more information in the "What risks can I expect from taking part in this study?" section.

If you choose to take part in this study, there is a risk that the study treatment may not be as good as usual treatments at shrinking or stabilizing your cancer.


There is also a risk that you could have side effects from the olaparib and/or temozolomide. These side effects may be worse and may be different than those you would get with the usual approach for uterine leiomyosarcoma.

Some of the most common side effects that the study doctors know about are:

- Anemia ("low red blood cell count"), which may require blood transfusion.
- Diarrhea, constipation, nausea and/or vomiting
- Difficulty sleeping
- Dizziness
- Hair loss
- Loss of appetite
- Muscle weakness
- Tiredness
- Trouble with memory

Olaparib, one of the study drugs, has rarely been associated with the development of acute myeloid leukemia, an aggressive and potentially incurable type of blood cancer, and myelodysplastic syndrome, a condition in which the bone marrow does not properly make blood cells and which can later develop into blood cancer. Based on other studies conducted with olaparib by itself, the risk of these conditions occurring appears to be less than 1.5%. The study doctors will monitor your bloodwork regularly for signs of these conditions.

There may be some risks that the study doctors do not yet know about.

#### **Benefits**

The researchers do not know how well the combination of olaparib and temozolomide could work against your type of cancer. It is unlikely that olaparib and temozolomide will work in everyone with your cancer or help you live longer. This study may help the study doctors learn things that may help other people in the future.

# If I decide to take part in this study, can I stop later?

Yes, you can decide to stop taking part in the study at any time.

If you decide to stop, let your study doctor know as soon as possible. It's important that you stop safely. If you stop, you can decide if you want to keep letting the study doctor know how you are doing.

Your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

# Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:


- Your health changes and the study is no longer in your best interest.
- New information becomes available and the study is no longer in your best interest.
- You do not follow the study rules.
- You become pregnant while on the study.
- The study is stopped by the Institutional Review Board (IRB), Food and Drug Administration (FDA), or study sponsor (National Cancer Institute [NCI]). The study sponsor is the organization who oversees the study.

It is important that you understand the information in the informed consent before making your decision. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or nurse.

## What is the purpose of this study?

The purpose of this study is to test the good and bad effects of olaparib in combination with temozolomide for the treatment of advanced uterine leiomyosarcoma. Olaparib and temozolomide could shrink your cancer, but could also cause side effects, which are described in the risks section below. The study doctors hope to learn if the study drug will be a safe and effective treatment for people with this type of cancer.

The olaparib and temozolomide combination has not been approved by the FDA to treat cancer. Olaparib and temozolomide are approved by the FDA to treat certain types of cancer when used individually, but the combination has not been approved for the treatment of any type of cancer. Temozolomide is sometimes used by itself to treat certain types of cancer, including uterine leiomyosarcoma.

We don't know if the combination of olaparib and temozolomide will work to treat cancer in people.

There will be about 22 people taking part in this study.

# What are the study groups?

In this study, you will receive both of the study drugs: olaparib and temozolomide. All patients receive the same treatment. Both olaparib and temozolomide will be taken orally. Olaparib is taken twice per day, and temozolomide is taken once per day. Both drugs are taken for the first 7 days of each 21-day cycle. In other words, you will take the treatment for one week and then have 2 weeks off before restarting the treatment again. You should not consume grapefruit juice or Seville oranges while taking olaparib and you should take temozolomide on an empty stomach.

You will not be able to get additional doses of olaparib and temozolomide. This treatment combination is not approved by the FDA for treatment of your disease.


## What exams, tests, and procedures are involved in this study?

Before you begin the study, your doctor will review the results of your exams, tests, and procedures. This helps your doctor decide if it is safe for you to take part in the study. If you join the study, you will have more exams, tests, and procedures to closely monitor your safety and health. Most of these are included in the usual care you would get even if you were not in a study.

Listed below are exams, tests, and procedures that need to be done as part of this study to monitor your safety and health, but may not be included in the usual care. We will use them to carefully follow the effects of the study treatment, including preventing and managing side effects.

These exams, tests, and procedures to monitor your safety and health include:

- Physical examinations and blood tests once every 3 weeks. For the first two cycles of treatment (first 6 weeks of treatment), a blood test will occur weekly. Some of these blood tests may be performed locally, at the discretion of your doctor. If you have been on study more than 2 years, a telephone or TeleHealth visit may be performed every other cycle, at the discretion of your doctor.
- A biopsy of your tumor before starting treatment and during the fourth week of the study. Imaging tests, such as CT scans, to help monitor the status of your cancer. These imaging tests will be performed approximately once every 6 weeks. For patients who continue beyond 12 cycles, MRI or CT imaging may be changed to once every 4 cycles (12 weeks) ± 3 days versus once every 6 weeks.

This study will use genetic tests that may identify changes in the genes in your tumor DNA and in the DNA of your normal cells. Your genes carry information about you and your family, from the color of your eyes to health conditions for which you may be at risk, including certain kinds of cancer.

Finding these changes would not affect your treatment in this study. However, they could affect your health in other ways. If there are changes found that could cause health problems, then your study doctor will discuss your options with you.

You will need to have biopsies for this study. A biopsy of a site of tumor will be performed twice. The first biopsy will be performed prior to starting the study treatment. The second biopsy will be performed during the fourth week of study treatment. The biopsy takes small pieces of cancer tissue from your body. This is like the biopsy you had to diagnose your cancer. In addition, you will need to have a blood sample taken before starting the study treatment. The biopsy and blood will be used to help the researchers understand which patients may benefit most from the study treatment and to evaluate whether the study treatment is working in the way it was intended to work. You and your study doctor will not get the results of this testing. If you


agree to take part in the study, you may need to sign a separate consent form for the study biopsy at the hospital or clinic where the biopsy is done.

A patient study calendar is attached at the end of this document. It shows how often blood sample collections, imaging tests, and biopsies will be done.

## What risks can I expect from taking part in this study?

#### **General Risks**

If you choose to take part in this study, there is a risk that the olaparib and temozolomide may not be as good as the usual approach at shrinking or stabilizing your cancer.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in certain future studies.

The olaparib and temozolomide combination used in this study could be very harmful to an unborn or newborn baby. There may be some risks that doctors do not yet know about. It is very important that you check with your study doctor about what types of birth control or pregnancy prevention you should use during the study and for 3 months after you have completed the study.

#### **Genetic Testing Risks**

The genetic tests used in this study will test your tumor and normal tissue for certain genetic changes. This study will specifically test for changes in certain genes that control how a cell repairs damage to DNA, including the following genes: BRCA1, BRCA2, ATM, ATR, ATRX, CHK1, CHK2, RAD51, PALB2, FANCA, and NBS1. If you have specific questions about what these genes are, ask your doctor. Changes found in your normal tissue may be passed down in families. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down.

Genetic tests of normal tissue can reveal information about you and also about your relatives. Your doctor will talk with you about what testing your normal tissue may mean for you and your family. He or she also may suggest that you talk with a genetics counselor to learn more. You or your insurance plan would have to pay for any genetic tests and/or visits to a genetic counselor done outside of this study.

#### **Biopsy Risks**

Common side effects of a biopsy are a small amount of bleeding at the time of the procedure, bruising, and pain at the biopsy site. Pain can be treated with regular pain medications. Rarely,


an infection, significant bleeding and injury to an internal organ could occur. You may sign a separate consent form for the study biopsy that describes these risks in more detail.

#### **Blood Draw Risks**

Blood draws for research may require an additional needle stick. Some of the risks from drawing blood from your arm may include pain, bruising, lightheadedness, and rarely, infection. Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

#### Side Effect Risks

The drugs used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood and let you know if changes occur that may affect your health.

There is also a risk that you could have other side effects from the study drugs.

Here are important things to know about side effects:

- 1. The study doctors do not know who will or will not have side effects.
- 2. Some side effects may go away soon, some may last a long time, and some may never go away.
- 3. Some side effects may make it hard for you to have children.
- 4. Some side effects may be mild. Other side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if there is a side effect.
- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.

This study is looking at a chemotherapy drug used to treat this type of cancer (temozolomide) plus a study drug not previously used in this cancer (olaparib). This different combination of drugs may increase your side effects compared to the individual drugs alone, or may cause new side effects.

#### **Drug Risks**

The tables below show the most common and most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.


#### Possible Side Effects of Olaparib (AZD2281; CAEPR Version 2.6, June 5, 2023)

#### COMMON, SOME MAY BE SERIOUS

In 100 people receiving olaparib (AZD2281), more than 20 and up to 100 may have:

- Anemia which may require blood transfusion
- Pain
- Diarrhea, nausea, vomiting
- Tiredness
- Loss of appetite

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving olaparib (AZD2281), from 4 to 20 may have:

- Bloating, constipation, heartburn
- Sores in the mouth which may cause difficulty swallowing
- Swelling of arms, legs
- Cold symptoms such as stuffy nose, sneezing, sore throat
- Infection which may cause painful and frequent urination
- Infection, especially when white blood cell count is low
- Dizziness, headache
- Changes in taste
- Cough, shortness of breath
- Rash

#### RARE, AND SERIOUS

In 100 people receiving olaparib (AZD2281), 3 or fewer may have:

- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Bruising, bleeding
- Cancer of bone marrow caused by chemotherapy
- Damage to the bone marrow (irreversible) which may cause infection, bleeding, may require transfusions
- Damage to the lungs which may cause shortness of breath
- Blood clot

## Possible Side Effects of Temozolomide (Table Version Date: May 23, 2017)

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Temozolomide, more than 20 and up to 100 may have:

- Constipation, nausea, vomiting, diarrhea
- Dizziness
- Muscle weakness, paralysis, difficulty walking
- Trouble with memory
- Tiredness
- Difficulty sleeping


#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Temozolomide, more than 20 and up to 100 may have:

• Hair loss

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Temozolomide, from 4 to 20 may have:

- Headache, seizure
- Infection, especially when white blood cell count is low
- Anemia which may cause tiredness
- Bruising, bleeding

#### RARE, AND SERIOUS

In 100 people receiving Temozolomide, 3 or fewer may have:

- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Cancer of bone marrow caused by chemotherapy
- Damage to the bone marrow (irreversible) which may cause infection, bleeding, may require blood transfusions
- Rash
- Severe skin rash with blisters and can involve inside of mouth and other parts of the body
- Liver damage which may cause yellowing of eyes and skin, swelling
- Cough, damage to the lungs which may cause shortness of breath

## **Additional Drug Risks**

The study drug could interact with other drugs. Your study doctor will give you a drug information handout and wallet card that lists these possible interactions. Share this information with your family members, caregivers, other health care providers, and pharmacists.

Rarely, there are problems getting enough supplies of the study drug. If that happens, your doctor will talk with you about your options.

#### **Imaging Risks**

The CT scans performed in this study will expose you to low amounts of radiation. Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. This type of radiation is called "background radiation." No one knows for sure whether exposure to these low amounts of radiation is harmful to your body. CT scans to monitor the status of your cancer will be done with similar frequency on this study as if you were receiving standard treatment for your cancer. However, 2-3 additional CT scans may be performed during the biopsy procedures. Each of these procedures will expose you to a very small amount of radiation (approximately 30 mSV) in addition to the amount that you might receive from your normal medical care. There may be an increase in the chances of your developing another cancer many years after this study. We estimate that this could happen in about 1 out of every 1000 people who get a very large amount of extra radiation. At this very low level, scientists are uncertain as to the actual risk from research and there may be no risk at all.


## What are my responsibilities in this study?

If you choose to take part in this study you will need to:

- Keep your study appointments.
- Tell your doctor about:
  - o all medications and supplements you are taking
  - o any side effects you are feeling
  - o any doctors' visits or hospital stays outside of this study
  - o if you have been or are currently in another research study.
- Write down in your medication diary when you take the study drug at home.

Do not get pregnant or breastfeed while taking part in this study. Tell your study doctor right away if you think that you have become pregnant during the study or within 3 months after your last dose of study drug.

## What are the costs of taking part in this study?

You and/or your insurance plan will need to pay for the costs of medical care you get as part of the study, just as you would if you were getting the usual care for your uterine leiomyosarcoma. This includes:

- the costs of tests, exams, procedures, and drugs that you get during the study to monitor your safety, and prevent and treat side effects.
- the cost of temozolomide
- the costs of getting temozolomide ready and giving it to you.
- your insurance co-pays and deductibles.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.

Ask your doctor or nurse for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You and/or your insurance provider will not have to pay for exams, tests, and procedures done for research purposes only or that are covered by the study. These include the two biopsy procedures performed as part of study participation. You or your insurance provider will also not have to pay for olaparib while you take part in this study. Temozolomide is listed on the National Comprehensive Cancer Network (NCCN) guidelines for the treatment of sarcoma. In most cases, the cost of temozolomide is expected to be covered by your insurance. However, if insurance is not willing to pay for temozolomide, and there is no other means to access the medication, you may not be able to participate in this study.

Taking part in this study may mean that you need to make more visits to the clinic or hospital than if you were getting the usual approach to treat your cancer. You may:


- Have more travel costs.
- Need to take more time off work.
- Have other additional personal costs.

You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

## What happens if I am injured because I took part in this study?

If you are injured as a result of taking part in this study and need medical treatment, please talk with your study doctor right away about your treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. Agreeing to take part in this study does not mean you give up these rights.

## Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

There are organizations that may look or receive copies of some of the information in at your study records. Your health information in the research database also may be shared with these organizations. They must keep your information private, unless required by law to give it to another group.

Some of these organizations are:

- The study sponsor and any company supporting the study now or in the future. This would include any organization helping the company with the study.
- The NCI Central IRB, which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The FDA and the groups it works with to review research


• The NCI and the groups it works with to review research.

In addition to storing data in the study database, data from studies that are publicly funded may also be shared broadly for future research with protections for your privacy. The goal of this data sharing is to make more research possible that may improve people's health. Your study records may be stored and shared for future use in public databases. However, your name and other personal information will not be used.

Some types of future research may include looking at your information and information from other patients to see who had side effects across many studies or comparing new study data with older study data. However, right now we don't know what research may be done in the future using your information. This means that:

- You will not be asked if you agree to take part in the specific future research studies using your health information.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

There are laws that protect your genetic information. However, there is a risk that someone could get access to your genetic information and identify you by name. In some cases, employers could use your genetic information to decide whether to hire or fire you. The study doctors believe the risk of this happening is very small. However, the risk may increase in the future as people find new ways of tracing information. For more information about the laws that protect you, ask your study doctor.

## Where can I get more information?

You may visit the NCI web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns you have about this study or to report side effects or injuries. Contact the study doctor (\*insert name of study doctor[s]\*) at (\*insert telephone number, and email address if appropriate\*).

For questions about your rights while in this study, call the (\*insert name of organization or center\*) Institutional Review Board at (\*insert telephone number\*).

# Optional studies that you can choose to take part in


This part of the consent form is about optional studies that you can choose to take part in. They are separate from the main study described above. These optional studies will not benefit your health. The researchers leading these optional studies hope the results will help other people with cancer in the future. The results will not be added to your medical records and you or your study doctor will not know the results.

Taking part in these optional studies is your choice. You can still take part in the main study even if you say "no" to any or all of these studies. There is no penalty for saying "no." You and your insurance company will not be billed for these optional studies. If you sign up for, but cannot complete any of these studies for any reason, you can still take part in the main study.

Circle your choice of "yes" or "no" for each of the following studies:

#### **Known future studies**

If you choose to take part in these optional studies, researchers will collect your tumor tissue as described below:

## Additional (3<sup>rd</sup>) Tumor Biopsy

The drugs that are used to treat cancer sometimes work for a period of time, but then stop working. In most cases, the reasons the drugs stop working are not known. The researchers suspect the cancer may change to develop "resistance" to the drugs in some way. In order to understand how to make the drugs work better, the researchers would like to take an additional tumor biopsy from patients who the drugs help initially, but then the cancer starts to get larger at a later time. The researchers will use this additional biopsy to study changes that have occurred in the tumor when it starts growing again. Not all patients will be asked to undergo this biopsy. Only patients whose tumor shrinks or who have stabilization of their cancer for more than 12 weeks and who then have a certain amount of growth in the cancer will be asked to undergo this biopsy. This biopsy is conducted while patients are still receiving the study treatment, but the cancer has started to grow only a small amount. The study doctors will notify you if you are appropriate for this test.

#### **Unknown future studies**

If you choose to take part in this optional study, any of your tumor tissue or blood samples left over from the genomic sequencing and other research tests specifically performed for this study will be stored. Storing samples for future studies is called "biobanking." The biobank is being run by the Nationwide Children's Hospital in Columbus, Ohio, and is supported by the NCI. Also, any health-related information, such as your response to cancer treatment, results of study tests, and medicines you took, will be stored for future use. Your genomic sequence will also be stored in a secure NIH database for future use. There is no limit on the length of time we will keep your samples and research information. The samples will be kept until they are used for research or destroyed. This is a publicly funded study. Samples from publicly funded studies are required to be shared as broadly as possible. However, we will protect your privacy. The goal of this is to make more research possible that may improve people's health.


The biobank is a public research resource. It has controlled access. This means that researchers who want to get samples and data from it must submit a specific research request. The request identifies who they are and what their planned research project is. Before getting the samples and data, the researchers must agree to keep the data private, only use it for their planned research project, and never use it to try to identify you.

Right now, we do not know what research may be done in the future using your tumor tissue and blood samples. This means that:

- You will not be asked if you agree to take part in the future research studies.
- You and your study doctor will not be told when or what type of research will be done.
- Future research studies may include genomic sequencing.
- You will not get reports or other information about any research that is done using your samples.

Unknown future research studies may include sequencing of all or part of your DNA. This is called genomic sequencing. Sequencing allows researchers to identify your genetic code. Changes in your genetic code may just be in your tumor tissue. These are called somatic changes. Changes may also be in your normal tissue and passed down through your family. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down. These are called germline changes.

If only tumor tissue is sequenced, we will not know if a genetic change in your tumor is also in your normal tissue. This is why sometimes both normal tissue and tumor tissue are sequenced. This helps researchers understand if a genetic change happened only in your cancer tissue, or in your normal tissue as well.

#### What is involved in this optional sample collection?

If you agree to take part, here is what will happen next:

- 1. A sample from the tissue that was collected prior to starting the study and during the fourth week of study participation will be sent to the biobank. A sample of tissue may be collected from an optional extra biopsy if the study drugs initially help but you then your tumor starts to get larger again. If you participate in this part of the study, the study doctors will tell you if the biopsy is appropriate for you. There is a chance you may not be appropriate for the biopsy and it will not be performed. The biopsy procedure is identical to the other biopsy procedures performed on the study as described above in the section "What exams, tests and procedures are involved in this study?"
- 2. Your samples will be stored in the biobank. There is no limit on the length of time we will keep your samples and research information. The samples will be kept until they are used for research or destroyed.
- 3. Researchers can only get samples from the biobank after their research has been approved by experts. Researchers will not be given your name or contact information.


4. Some of your genetic and health information may be placed in central databases for researchers to use. The databases will not include your name or contact information.

#### What are the risks in this optional sample collection?

- The most common risks related to a biopsy are a small amount of bleeding at the time of the procedure, bruising, and pain at the biopsy site. Pain can be treated with regular pain medications. Rarely, an infection, significant bleeding, or damage to an organ can occur.
- Your medical and genetic information is unique to you. There is a risk that someone
  outside of the research study could get access to your study records or trace information
  in a database back to you. They could use that information in a way that could harm you.
  Researchers believe the chance that someone could access and misuse your information is
  very small. However, the risk may increase in the future as people find new ways of
  tracing information.
- In some cases, this information could be used to make it harder for you to get or keep a job and get or keep health insurance.

#### How will information about me be kept private?

Your privacy is very important to the study researchers and biobank. They will make every effort to protect it. Here are just a few of the steps they will take:

- 1. They will remove identifiers, such as your initials, from your sample and information. They will replace them with a code number. There will be a master list linking the code numbers to names, but they will keep it separate from the samples and information.
- 2. Researchers who study your samples and information will not know who you are. They also must agree that they will not try to find out who you are.
- 3. Your personal information will not be given to anyone unless it is required by law.
- 4. If research results are published, your name and other personal information will not be used.

#### What are the benefits to taking part in this optional sample collection?

You will not benefit from taking part. The researchers, using the samples from you and others, might make discoveries that could help people in the future.

#### Are there any costs or payments to this optional sample collection?

There are no costs to you or your insurance. You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

#### What if I change my mind about this optional sample collection?

If you decide you no longer want your samples to be used, you can call the study doctor, Brian Van Tine, M.D., Ph.D., at 314-747-3096.


## What if I have questions about this optional sample collection?

If you have questions about the use of your samples for research, contact the study doctor, Brian Van Tine, M.D., Ph.D., at 314-747-3096.

Please circle your answer below to show if you would or would not like to take part in each optional study:

# Samples for known future studies: Additional (3<sup>rd</sup>) Tumor Biopsy

<u>Please circle your answer</u>: I choose to permit an additional tumor biopsy if the study treatment appears to help me, but my cancer later starts to grow.

YES NO

#### Samples for unknown future studies:

I agree that my samples and related health information may be kept in a biobank for use in future health research.

YES NO

This is the end of the section about optional studies.

## My signature agreeing to take part in the study

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed and dated copy of this form. I agree to take part in the main study. I also agree to take part in any additional studies where I circled "yes".

#### Participant's signature

Date of signature

#### Signature of person(s) conducting the informed consent discussion


Date of signature


## **Attachment 1: Study Calendar**

| | | Cycle 1 | | | Cycle 2 | | | Cycle 3+ | | | Pre- | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre-study <sup>G</sup> | Wk | Wk<br>2 | Wk<br>3 | Wk<br>4 <sup>K</sup> | Wk<br>5 | Wk<br>6 | Wk<br>7 <sup>K</sup> | Wk<br>8 | Wk<br>9 | Progression | Off Study <sup>D</sup> |
| Olaparib <sup>A</sup> | | 1<br>X <sup>A</sup> | 2 | 3 | X <sup>A</sup> | 3 | 0 | XA | 0 | 9 | | |
| Temozolomide <sup>B</sup> | | $X^{B}$ | | | $X^{B}$ | | | $X^{B}$ | | | | |
| Pre-study procedures including informed consent, demographics, medical history, and height measurement | Х | | | | | | | | | | | |
| Physical exam <sup>L</sup> ,<br>concurrent meds, vital<br>signs <sup>M</sup> , and general<br>well-being | X | X <sup>I</sup> | | | X <sup>I</sup> | | | X <sup>I</sup> | | | | X |
| Weight | X | X <sup>I</sup> | | | X <sup>I</sup> | | | X <sup>I</sup> | | | | X |
| Blood draw for<br>complete blood count<br>and general health<br>status | X | X <sup>I</sup> | $X^{J}$ | X <sup>J</sup> | X <sup>I</sup> | $X^{J}$ | $X^{J}$ | X <sup>I</sup> | | $X^{J}$ | | X |
| Blood test to measure<br>how well your blood<br>clots | X | X <sup>I</sup> | | | X <sup>I</sup> | | | X <sup>I</sup> | | | | X |
| ECG <sup>H</sup> | X | | | | | | | | | | | X |
| CT/MRI Imaging to<br>monitor disease<br>status <sup>E</sup> | X | | | | | | X | | | | | X |
| Pregnancy test <sup>C</sup> | X | X | | | X | | | X | | | | X |
| Tumor Biopsy <sup>F</sup> | X | | | | X | | | | | | | |
| Optional Tumor<br>Biopsy for Selected<br>Patients | | | | | | | | | | | X | |
| Blood Collection for<br>Research | X | | | | | | | | | | | |

- A: Olaparib: 200 mg by mouth, twice a day, on days 1-7 of a 21-day cycle. Dosing window of ± 2 days at the start of each cycle is allowed; however, both agents must begin dosing on the same day.
- B: Temozolomide:  $75 \text{ mg/m}^2$  by mouth, once a day, on days 1-7 of a 21-day cycle. Dose is based on weight at screening. Dosing window of  $\pm$  2 days at the start of each cycle is allowed; however both agents must begin dosing on the same day.
- C: Serum or urine pregnancy test (for women of childbearing potential) must be completed within 14 days of the start of study treatment, on Day 1 of the study prior to commencing treatment, at each subsequent visit during study treatment, and at the follow up visit.
- D: Off-study evaluations must be performed within 21 days of the last dose of study drug.
- E: MRI or CT imaging to evaluate response and disease status is performed every 2 cycles (6 weeks) ± 3 days. For patients who continue beyond 12 cycles, MRI or CT imaging may be changed to once every 4 cycles (12 weeks) ± 3 days versus once every 6 weeks.
- F: Pre-study biopsy is performed within 14 days of Cycle 1 Day 1. On study biopsy is performed on day 3-5 of Cycle 2. If the start of Cycle 2 is delayed, the biopsy may be delayed accordingly to match Day 3-5 based upon the actual day of dosing reinitiation.
- G: All pre-study screening procedures must be completed within 14 days of C1D1. Informed consent must be completed within 21 days of C1D1. Blood testing and imaging obtained as part of standard of care and which falls within this timeframe and otherwise meets protocol specifications need not be repeated.
- H: A 12-lead ECG is performed at screening and end-of-study. Additional EKGs are performed as clinically indicated.
- Assessments may be performed up to 3 days prior to initiating treatment for a new cycle. Local laboratory testing is acceptable.
- J: Between cycle safety assessments may be performed ± 3 days from scheduled date. Local laboratory testing is acceptable.
- K: New cycle may begin  $\pm 2$  days from scheduled date.
- L: A complete physical exam is performed at screening and end-of-study. A limited, symptom based, physical exam is performed at other timepoints. If you have been on the study more than 2 years, a telephone or TeleHealth visit may be performed every other cycle, at the discretion of your doctor.
- M: Vital signs includes measurement of temperature, heart rate, blood pressure, respiratory rate, and oxygen saturation (pulse oximetry).
